CLINICAL TRIAL: NCT06649539
Title: Efficacy of a Step-wise Protocol in Optimizing CCH Outcomes in Men With Peyronie's Disease
Brief Title: Delayed Dose Collagenase Clostridium Histolyticum (CCH) Protocol for Men With Peyronie's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charitable Union for the Research and Education of Peyronie's Disease (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Landon Trost, Principal Investigator, MD, Charitable Union for the Research and Education of Peyronie's Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUREPD120
Record Dates: First submitted 2024-10-12; First posted 2024-10-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Peyronie Disease
Keywords: collagenase clostridium histolyticum; curvature; Restorex; Xiaflex; traction; salvage
MeSH Terms: conditions — Penile Induration | interventions — Microbial Collagenase; Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: prospective, single-blinded clinical trial
Masking Description: Investigators will be blinded to baseline curvature measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Primary Cohort (Experimental): Men would receive 4 series of CCH injections:
  * Administered on back-to-back days
  * 0.9 mg administered with each series, diluted to 0.8 mL
  * Mild in-office modeling performed on treatment day 2 of each series
  * Wraps applied 2-4 full-time and 2-4 part-time days
  * Sildenafil 25 mg nightly and Restorex beginning treatment day 2 (sildenafil) or 3 (Restorex - 30 min/day) until 6 weeks after final injection of the final series.
  Note that men may stop sooner if they are satisfied before completing the 4 series. If the patient is not satisfied with outcomes by the end of the 4th series, they would be permitted to enter the 'salvage' phase of the treatment protocol.
  * Performed 9-12 months after the 4th series of injections.
  * The technique would incorporate more aggressive, in-office modeling.
  * Men would receive up to two additional series per this protocol.
  Interventions: Drug: Collagenase Clostridium Histolyticum; Device: RestoreX; Drug: Sildenafil

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum — 4 Series given to each participant, 6 weeks apart. Medication administered on back-to-back days. If failing to achieve an adequate response, men may receive up to 2 additional series 9-12 months after the 4th series.
  Total of 0.9 mg administered with each series, diluted to 0.8 mL
  Other Names: Xiaflex; CCH
Device: RestoreX — Restorex initiated beginning on post-injection day 3 or as soon as tolerated - 30 min daily, continuing until 6 weeks after final injection of the final CCH series.
Drug: Sildenafil — Men will be prescribed sildenafil 25 mg nightly beginning treatment day 2 until 6 weeks after final injection of the final series.
  Other Names: Viagra

SUMMARY:
Our team has previously demonstrated efficacy in performing a novel collagenase Clostridium histolyticum (CCH) injection protocol in men who previously failed to achieve a response to an initial 4 series of CCH.

The objective of the current study is to evaluate a protocol that incorporates limited in-office modeling for up to 4 series, followed by up to 2 additional salvage series to determine safety and efficacy compared to historical data.

Participants will receive up to 4 series of CCH injections using our previously published protocol, with mild in-office modeling. CCH injections are given on back-to back days, after which they are counseled to utilize Restorex and sildenafil daily, as instructed. Patients will undergo mild in-office modeling on day 2.

The sexual partners of study participants will also be invited to enroll in the study and will complete non-validated questionnaires detailing their level of support for the patient's treatment.

DETAILED DESCRIPTION:
The current study would prospectively follow 40 men through the following treatment protocol:

* Men would receive 4 series of CCH injections according to the protocol below, which represents a modified version of our most recently published technique.13

  * Medication administered on back-to-back days
  * Total of 0.9 mg administered with each series, diluted to 0.8 mL
  * Mild in-office modeling performed on treatment day 2 of each series
  * Wraps performed ranging from 2-4 full-time and 2-4 part-time days to minimize bruising
  * Sildenafil 25 mg nightly beginning treatment day 2 until 6 weeks after final injection of the final series.
  * Restorex initiated beginning on post-injection day 3 or as soon as tolerated - 30 min daily, continuing until 6 weeks after final injection of the final series.
* Note that men may stop sooner if they are satisfied before completing the 4 series.
* If the patient is not satisfied with outcomes by the end of the 4th series, they would be permitted to enter the 'salvage' phase of the treatment protocol.

  * This would be performed 9-12 months after the 4th series of injections.
  * The technique would be similar to the one noted above with the exception of more aggressive in-office modeling as described in our prior publication and per our ongoing randomized trial.
  * The men would receive up to two additional series per this protocol for a maximum number of cycles being 6 in total.

At the time of initial enrollment, partners of study participants will be invited to enroll in the study and will be administered non-validated questionnaires designed to assess the partner's overall support for the ongoing treatment protocol.

Assessments and study questionnaires will be administered at baseline, with the 1st injection of each series, 6 weeks after completing the 4th series of CCH injections, and 1 year after completion of the final series of CCH injections.

ELIGIBILITY:
Inclusion Criteria:

* Men with Peyronie's Disease
* Older than 18 years old
* Curvature ≥30 degrees
* Ability to achieve an erection satisfactory for intercourse with or without phosphodiesterase-5 (PDE5) inhibitors
* The patient exhibits a palpable plaque consistent with Peyronie's Disease
* For partners, the only inclusion criteria is being willing to complete a questionnaire

Exclusion Criteria:

* Prior surgical treatment on the penis (other than circumcision)
* Prior treatment with CCH injections
* Any contraindications to CCH - as determined by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Penile Curvature | 1 year
  Compare penile curvature between baseline and post-treatment in men 1 year after completing the final injection series. A goniometer (protractor) will be used to measure from the penile angulation during a full erection in two planes (dorsal/ventral and lateral). Measurements will be in degrees.
Penile Length | 1 year
  Compare penile length between baseline and post-treatment in men 1 year after completing the final injection series. Measurements will be performed using a ruler, with measurements obtained from the pubic symphysis to the corona of the glans penis (measured in cm).

SECONDARY OUTCOMES:
Penile curvature compared to more aggressive technique | 1 year
  Compare curvature outcomes to our historical series of men treated up-front with the more aggressive technique. This will be done using a goniometer (protractor) with a full erection and measured in two planes (dorsal/ventral and lateral). The curvature will be measured using degrees.
Penile curvature compared to our current salvage approach for CCH | 1 year
  Compare curvature changes to those in our ongoing randomized, controlled trial (NCT05108558) evaluating the salvage approach in men who previously failed 6-8 CCH injections. This will be done using a goniometer (protractor) with a full erection and measured in two planes (dorsal/ventral and lateral). The curvature will be measured using degrees.
Adverse Events | 1 year
  Report subjectively noted adverse events (AE) at 1 year following the final injection series. Patients will be able to write-in specific adverse events, and absolute occurrences of each of the written responses will be summed and reported.
Partner Support | 1 year
  Evaluate partner support as a predictor of whether the patient continues with treatment. Support will be assessed using a non-validated question, "How supportive are you of your partner's decision to undergo Xiaflex treatments?" This will be measured using the selectable options: Very Supportive, Somewhat Supportive, Neutral, Somewhat Unsupportive, and Very Unsupportive.
Compliance with Therapy - Penile Curvature | 1 year
  Evaluate compliance with therapy as a predictor of penile curvature improvements during the study. A daily diary will be maintained by the patient to track actual device utilization. Patients will record how many minutes that they used the device daily. This information will be used to try to correlate penile curvature outcomes with actual device utilization.
Satisfaction with therapy | 1 year
  Report patient-outcome measures related to satisfaction with therapy. This measure will be evaluated using a non-standardized question, "How would you rate your overall satisfaction with Xiaflex?" Patients will be able to select from the following responses: Very Satisfied, Somewhat Satisfied, Neither Satisfied nor Dissatisfied, Somewhat Dissatisfied, Very Dissatisfied.
Penile length compared to more aggressive technique | 1 year
  Compare penile length changes to our historical series of men treated up-front with the more aggressive technique. Measurements will be performed using a ruler, with measurements obtained from the pubic symphysis to the corona of the glans penis (measured in cm).
Penile length compared to our current salvage approach for CCH | 1 year
  Compare penile length changes to our ongoing randomized, controlled trial (NCT05108558) evaluating the salvage approach in men who previously failed 6-8 CCH injections. Measurements will be performed using a ruler, with measurements obtained from the pubic symphysis to the corona of the glans penis (measured in cm).
Compliance with Therapy - Penile Length | 1 year
  Evaluate compliance with therapy as a predictor of penile length changes during the study. A daily diary will be maintained by the patient to track actual device utilization. Patients will record how many minutes that they used the device daily. This information will be used to try to correlate penile length outcomes with actual device utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Landon Trost, MD, Principal Investigator — Charitable Union for the Research and Education of Peyronie's Disease
Locations (1):
- Male Fertility and Peyronie's Clinic, Orem, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen HMT, Anaissie J, DeLay KJ, Yafi FA, Sikka SC, Hellstrom WJG. Safety and Efficacy of Collagenase Clostridium histolyticum in the Treatment of Acute-Phase Peyronie's Disease. J Sex Med. 2017 Oct;14(10):1220-1225. doi: 10.1016/j.jsxm.2017.08.008. Epub 2017 Sep 2. PMID 28874331
- [Background] Larson H, Warner J, Savage J, Kohler T, Ziegelmann M, Trost L. Changes in Point of Maximal Curvature During Collagenase Clostridium Histolyticum Injections for Peyronie's Disease. Urology. 2024 Feb;184:122-127. doi: 10.1016/j.urology.2023.11.024. Epub 2023 Dec 6. PMID 38061610
- [Background] Gelbard M, Lipshultz LI, Tursi J, Smith T, Kaufman G, Levine LA. Phase 2b study of the clinical efficacy and safety of collagenase Clostridium histolyticum in patients with Peyronie disease. J Urol. 2012 Jun;187(6):2268-74. doi: 10.1016/j.juro.2012.01.032. Epub 2012 Apr 13. PMID 22503048
- [Background] Alom M, Sharma KL, Toussi A, Kohler T, Trost L. Efficacy of Combined Collagenase Clostridium histolyticum and RestoreX Penile Traction Therapy in Men with Peyronie's Disease. J Sex Med. 2019 Jun;16(6):891-900. doi: 10.1016/j.jsxm.2019.03.007. Epub 2019 Apr 5. PMID 30956106
- [Background] Ziegelmann MJ, Viers BR, Montgomery BD, Westerman ME, Savage JB, Trost LW. Self-reported Clinical Meaningfulness Early in the Treatment Course Predicts Objective Outcomes in Men Undergoing Collagenase Clostridium histolyticum Injections for Peyronie Disease. Urology. 2017 Aug;106:107-112. doi: 10.1016/j.urology.2017.04.045. Epub 2017 May 5. PMID 28483591
- [Background] Ziegelmann MJ, Viers BR, McAlvany KL, Bailey GC, Savage JB, Trost LW. Restoration of Penile Function and Patient Satisfaction with Intralesional Collagenase Clostridium Histolyticum Injection for Peyronie's Disease. J Urol. 2016 Apr;195(4 Pt 1):1051-6. doi: 10.1016/j.juro.2015.10.065. Epub 2015 Oct 23. PMID 26476353
- [Background] Alom M, Meng Y, Sharma KL, Savage J, Kohler T, Trost L. Safety and Efficacy of Collagenase Clostridium Histolyticum in Peyronie's Disease Men With Ventral Curvatures. Urology. 2019 Jul;129:119-125. doi: 10.1016/j.urology.2019.01.055. Epub 2019 Mar 22. PMID 30910455